CLINICAL TRIAL: NCT00456703
Title: Safety and Efficacy of Restricted Fluid Regimen in Open Abdominal Bowel Surgery
Brief Title: Restricted Fluid Regimen in Open Abdominal Bowel Surgery
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of funding
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Balachundhar Subramaniam, Associate Professor of Anaesthesia, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2006P000144
Record Dates: First submitted 2007-04-04; First posted 2007-04-05 (Estimated); Last update posted 2017-03-06 (Actual); Status verified 2017-03

CONDITIONS: Bowel Surgery
Keywords: fluids,; restriction,; infection,; bowel surgery,; open abdominal
MeSH Terms: conditions — Infections

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- restriction (Active Comparator): In this group, the fluids will be restricted compared to a standard procedure
  Interventions: Other: intraoperative fluid management; Other: fluid restriction

INTERVENTIONS:
Other: intraoperative fluid management — fluid restriction
Other: fluid restriction — restriction of fluids

SUMMARY:
Liberal intravenous fluid resuscitation during open abdominal surgery may predispose the patients to multiorgan dysfunction, prolong hospital stay and increase postoperative morbidity. The main aim of the study is to assess the safety and feasibility of restricted fluid regimen in open abdominal bowel surgery.

DETAILED DESCRIPTION:
This is a randomized, prospective controlled trial in patients (ASA I-III) undergoing open abdominal surgical procedures in a single center. This study will be done in two phases. The first phase is designed to evaluate and prove the safety of restricted fluid regimens in maintaining tissue perfusion using a central venous oximetric catheter and arterial blood gas analysis. In the second phase of the study, we plan to mimic the usual clinical practice without the central venous oximetric catheter and arterial lines (invasive monitors) and the postoperative total morbidity will be compared between the liberal and restricted fluid regimens.

In the first phase of the study, 90 patients coming in for open bowel surgery will be randomized to three groups using a random number generator. All patients will receive a standard bowel prep regimen (Go-Lyte-half a liter the night before surgery). Group A will receive current standard of care (liberal fluid therapy), Group B and C will receive restricted fluid regimens. All patients will receive 500 cc of intravenous fluids (lactated ringers in Group A and B, 6% hetastarch in Group C) in the preoperative holding area to correct preoperative fluid deficits due to fasting and bowel preparation. Patients younger than 18 years, ASA IV or V, pregnant patients, those with coagulopathy, renal insufficiency, unstable angina, unstable congestive heart failure, and those with contraindication to central venous pressure catheter insertion will be excluded from the study.

After instituting anesthesia monitors, patients will be anesthetized with a standard anesthetic regimen. An arterial line and a central venous catheter with oximetric capability will be inserted in all three groups. A baseline blood gas will be drawn to note the base excess, lactate levels and the hematocrit at the start of surgery. Parameters like heart rate, blood pressure, central venous pressure, mixed venous oxygen saturation and arterial oxygen saturation and urine output will be continuously monitored. Both the regimens will be started in the operating room and continued into the postoperative period until they resume their oral intake. Patients in the liberal group will receive (10ml/kg/hr) the current standard of care for bowel surgery whereas those in the restricted group will receive 4ml/kg/hour. Post induction hemodynamic instability will be treated with ephedrine and phenylephrine at the discretion of the anesthesiologist in charge.

Intraoperative treatment of tachycardia, hypotension in both the groups will be treated using a standard fluid regimen algorithm (appendix A). All patients will receive the same postoperative fluid regimens as the current standard of care. Postoperative morbidity evaluation (appendix B) will be done at patient's discharge from the hospital. The data entry will be prospectively done during their hospital stay. The accuracy of the data will be checked by one of the study investigators.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status I-III patients coming in for open abdominal bowel surgery

Exclusion Criteria:

* Coagulopathy,
* Pregnancy,
* Renal insufficiency,
* Contraindications for placing a central line,
* ASA IV and V,
* Age less than 18years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-07; Primary Completion 2009-07 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
mixed venous oxygen saturation, acid bases, hemodynamics | intraoperative period

SECONDARY OUTCOMES:
Wound infection and length of hospital stay | during the hospital admission

CONTACTS AND LOCATIONS:
Overall Officials: Balachundhar Subramaniam, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

REFERENCES:
- [Background] Nisanevich V, Felsenstein I, Almogy G, Weissman C, Einav S, Matot I. Effect of intraoperative fluid management on outcome after intraabdominal surgery. Anesthesiology. 2005 Jul;103(1):25-32. doi: 10.1097/00000542-200507000-00008. PMID 15983453
- [Background] Rivers E, Nguyen B, Havstad S, Ressler J, Muzzin A, Knoblich B, Peterson E, Tomlanovich M; Early Goal-Directed Therapy Collaborative Group. Early goal-directed therapy in the treatment of severe sepsis and septic shock. N Engl J Med. 2001 Nov 8;345(19):1368-77. doi: 10.1056/NEJMoa010307. PMID 11794169